CLINICAL TRIAL: NCT00812006
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Crossover Trial to Evaluate the Efficacy and Tolerability of Rizatriptan 10 mg ODT for the Treatment of Acute Migraine in Patients on Topiramate for Migraine Prophylaxis
Brief Title: A Study of Rizatriptan for the Treatment of Acute Migraine in Patients on Topiramate for Migraine Prophylaxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-085; 2008_597
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Results first posted 2011-01-27 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Treatment Sequence A: rizatriptan, rizatriptan, placebo
  Interventions: Drug: rizatriptan benzoate; Drug: Comparator: placebo
- B (Experimental): Sequence B: rizatriptan, placebo, rizatriptan
  Interventions: Drug: rizatriptan benzoate; Drug: Comparator: placebo
- C (Experimental): Sequence C: placebo, rizatriptan, rizatriptan
  Interventions: Drug: rizatriptan benzoate; Drug: Comparator: placebo

INTERVENTIONS:
Drug: rizatriptan benzoate — rizatriptan 10 mg Orally Disintegrating Tablet (ODT) orally for a moderate or severe migraine attack
  Other Names: Maxalt
Drug: Comparator: placebo — Placebo to rizatriptan 10 mg ODT orally for a moderate or severe migraine attack

SUMMARY:
This study will provide additional efficacy data for rizatriptan when used for an acute migraine attack in patients already taking topiramate for migraine prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of migraine with or without aura for more than one year, with between 2 and 8 moderate to severe attacks per month
* Patient is currently taking at least 50 mg topiramate daily for migraine prophylaxis
* Patient can distinguish between migraine and other types of headache
* Patient agrees to remain abstinent or use effective birth control during the study

Exclusion Criteria:

* Patient is pregnant or breast-feeding
* Patient has a history of mostly mild migraines or migraines that resolve within 2 hours
* Patient has more than 15 headache-days per month or has taken medication for acute headache on more than 10 days per month in the 3 months prior to screening.
* Patient was > 50 years old at age of migraine onset
* Patient has history of heart disease
* Patient has uncontrolled hypertension
* Patient has had cancer within 5 years of screening (excepting certain skin and cervical cancers)
* Patient has started taking Selective Serotonin Reuptake Inhibitors (SSRIs) or Serotonin-Norepinephrine Reuptake Inhibitors (SNRIs) or has changed doses within 3 months of screening
* Patient is taking more than one other migraine prophylactic medication
* Patient has repeatedly failed to respond to or tolerate rizatriptan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-03-24 (Actual); Primary Completion 2009-10-22 (Actual); Study Completion 2009-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seeburger JL, Cady RK, Winner P, MacGregor A, Valade D, Ge Y, Zhang Y, Hustad CM, Strickler N, Schaefer E, Connor KM, Ho TW. Rizatriptan for treatment of acute migraine in patients taking topiramate for migraine prophylaxis. Headache. 2012 Jan;52(1):57-67. doi: 10.1111/j.1526-4610.2011.02027.x. Epub 2011 Nov 11. PMID 22078129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 26 March 2009; Last Patient Last Visit: 22 October 2009.
  17 Outpatient centers worldwide (10 United States; 2 Canada; 2 Spain, 2 Italy; 1 France)
Pre-assignment Details: Participants were assessed, using the protocol inclusion and exclusion criteria, at Visit 1, and if eligible,
  were randomized at the same visit.
Groups:
- Rizatriptan / Rizatriptan / Placebo: First migraine treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); second migraine treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); third migraine treated with Placebo
- Rizatriptan / Placebo / Rizatriptan: First migraine treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); second migraine treated with Placebo; third migraine treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT)
- Placebo / Rizatriptan / Rizatriptan: First migraine treated with Placebo; second migraine treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); third migraine treated with Rizatriptan 10 mg Orally Disintegrating Tablet (ODT)
Period: Overall Study
Arm/Group | Rizatriptan / Rizatriptan / Placebo | Rizatriptan / Placebo / Rizatriptan | Placebo / Rizatriptan / Rizatriptan
Started | 36 | 36 | 36
Completed | 30 | 33 | 30
Not Completed | 6 | 3 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Lack of Qualifying Event | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rizatriptan / Rizatriptan / Placebo | Rizatriptan / Placebo / Rizatriptan | Placebo / Rizatriptan / Rizatriptan | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (12.0) | 43.9 (10.8) | 40.0 (11.6) | 44.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 34 | 99
  Male | 4 | 3 | 2 | 9
Ethnicity Origin [Number; unit: participants]
  Black | 0 | 1 | 0 | 1
  White | 36 | 35 | 36 | 107
Racial Origin [Number; unit: participants]
  Hispanic or Latino | 11 | 9 | 10 | 30
  Not Hispanic or Latino | 25 | 27 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief (PR)
Description: Pain severity was rated by the participants in a paper diary. Pain severity rating scale : 0 (no pain), 1 (mild pain), 2 (moderate pain), or 3 (severe pain). Pain relief (PR) is defined as a reduction in headache severity from Grade 3/2 at baseline to Grade 1/0 post dose.
Time Frame: 2 hours post dose
Population: Full Analysis Set, which included all randomized participants who had at least one evaluable attack. To be considered an evaluable attack, the participant must have administered study treatment for this attack and have both a baseline severity measurement and at least one post-dose efficacy measurement at or prior to the 2-hour time point.
Measure: Number; unit: Attacks
Groups:
- Rizatriptan: Rizatriptan 10 mg. Patients who treated at least one attack, that was intended to be treated with rizatriptan 10 mg (excluding sponsor-provided rescue), were included. Although a patient may have treated twice with rizatriptan 10 mg, the patient was counted only once for the rizatriptan group.
- Placebo: Placebo. Patients who treated one attack, that was intended to be treated with placebo, were included. One patient who treated an attack with placebo within 48 hours of the previous attack was excluded from the placebo group.
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 99 | 93
Attacks
  Resulting in PR at 2 hours post dose | 105 | 21
  Not resulting in PR at 2 hours post dose | 88 | 72
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model; An unstructured covariance matrix was used to model the correlation among repeated measurements within a patient

2. Secondary Outcome: Sustained Pain Relief (SPR)
Description: 24-hour sustained pain relief (defined as pain relief at 2 hours post dose, with no administration of any rescue medication and with no occurrence of a moderate/severe headache during the respective period after dosing with the blinded study medication.
Time Frame: 2 - 24 hours post dose
Population: Full Analysis Set, which included all randomized participants who had at least one evaluable attack. To be considered an evaluable attack, the attack must have met the FAS criteria for PR at 2 hours post-dose, and from 2-24 hours the participant either answered 24-hour headache recurrence question or didn't have PR at any time or took rescue.
Measure: Number; unit: Attacks
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 99 | 93
Attacks
  Resulting in SPR 2-24 hours post dose | 67 | 12
  Not resulting in SPR 2-24 hours post dose | 126 | 81
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model — Nominal p-value was adjusted under Benjamini and Hochberg's false discovery rate procedure for the multiple secondary endpoints at α=0.1 significance level; A compound-symmetry covariance matrix was used to model the correlation among repeated measurements within a patient, due to a convergence issue

3. Secondary Outcome: Pain Freedom (PF)
Description: Headache pain severity, relative to the administration of study medication, was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild pain), 2 (moderate pain), or 3 (severe pain). Pain freedom (PF) is defined as a reduction in headache severity from Grade 3/2 at baseline to Grade 0 (no pain) post dose.
Time Frame: 2 hours post dose
Population: as for outcome 1
Measure: Number; unit: Attacks
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 99 | 93
Attacks
  Resulting in PF 2 hours post dose | 74 | 9
  Not resulting in PF 2 hours post dose | 119 | 84
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model — [p-value comment as in outcome 2, analysis 1]; An unstructured covariance matrix was used to model the correlation among repeated measurements within a patient

4. Secondary Outcome: Normal Rating of Functional Disability (NRFD)
Description: Level of functional disability was assessed on a paper diary by the participants. Level of functional disability was rated as: normal, mildly impaired, severely impaired, or unable to do activities, requires bedrest. Functional disability ratings was dichotomized to Normal and Not Normal (mildly impaired, severely impaired, or unable to do activities, requires bedrest) for analysis.
Time Frame: 2 hours post dose
Population: as for outcome 1
Measure: Number; unit: Attacks
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 99 | 93
Attacks
  Resulting in NRFD at 2 hours post dose | 85 | 16
  Not resulting in NRFD at 2 hours post dose | 108 | 77
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model — Nominal p-value was adjusted under Benjamini and Hochberg's falsediscovery rate procedure for the multiple secondary endpoints at α=0.1 significance level; An unstructured covariance matrix was used to model the correlation among repeated measurements within a patient

5. Secondary Outcome: Treatment Satisfaction (TS)
Description: Patient satisfaction was assessed on a paper diary by the participants. Level of satisfaction was rated as: completely satisfied, very satisfied, somewhat satisfied, neither satisfied nor dissatisfied, somewhat dissatisfied, very dissatisfied, or completely dissatisfied. The overall 24-hour assessment of study medication was dichotomized to Satisfaction (completely satisfied, very satisfied, somewhat satisfied) and Non-satisfaction (neither satisfied nor dissatisfied, somewhat dissatisfied, very dissatisfied, or completely dissatisfied) for analysis.
Time Frame: 24 hours post dose
Population: Full Analysis Set, which included all randomized participants who had at least one evaluable attack. To be considered an evaluable attack, the participant must have administered study treatment for this attack and have both a baseline severity measurement and post-dose satisfaction measurement at the 24-hour time point.
Measure: Number; unit: Attacks
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 99 | 93
Attacks
  Resulting in TS at 24 hours post dose | 117 | 31
  Not resulting in TS at 24 hours post dose | 76 | 62
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; Test type: Superiority or Other; p < 0.001, Generalized Linear Mixed Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected up to 14 days after each qualified migraine headache attack that was treated with study medication.
Description: Adverse experiences were reported by the patient on a paper diary.
  Adverse events occurring within 14 days of administration of rizatriptan (including sponsor-provided rescue) are attributed to rizatriptan group, even if placebo was administered more recently
Groups:
- Rizatriptan: Rizatriptan 10 mg. Patients who treated at least one attack with rizatriptan 10 mg (including sponsor-provided rescue) were included. Although a patient may have treated twice with rizatriptan 10 mg, the patient was counted only once for the rizatriptan group. Adverse events occurring within 14 days of any administration of rizatriptan (including sponsor-provided rescue) were attributed to rizatriptan group, even if placebo was administered more recently.
  It is possible for one patient to be counted twice (once in each treatment group).
  The number of randomized patients is 108, out of which, 101 took at least one dose of rizatriptan (including sponsor-provided rescue), and 94 took placebo.
- Placebo: Placebo. Patients who treated an attack with placebo were included. Adverse events occurring within 14 days of administration of placebo, but not within 14 days of any administration of rizatriptan (including sponsor-provided rescue), were attributed to placebo group.
  It is possible for one patient to be counted twice (once in each treatment group).
  The number of randomized patients is 108, out of which, 101 took at least one dose of rizatriptan (including sponsor-provided rescue), and 94 took placebo.
Arm/Group | Rizatriptan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/94
Other Adverse Events (participants affected / at risk) | 16/101 | 3/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan (N=101) | Placebo (N=94)
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Temperature intolerance (General disorders) | 1 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Allodynia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Hypersomnia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Peripheral paralysis (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 6 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.